CLINICAL TRIAL: NCT04998279
Title: Intrauterine Infusion of Granulocyte Colony Stimulating Factor and Reproductive Outcomes in Infertile Women with History of Recurrent Implantation Failure
Brief Title: Intrauterine Infusion of GCSF and Reproductive Outcomes in Infertile Women with History of RIF
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Islam Tarek Elkhateb, principle investigator, Cairo University
Other Study IDs: 2464949
Record Dates: First submitted 2021-07-26; First posted 2021-08-10 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Recurrent Implantation Failure; Granulocyte Colony-Stimulating Factor; Infertility
MeSH Terms: conditions — Infertility | interventions — Granulocyte Colony-Stimulating Factor; Filgrastim

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Intervention group
  Interventions: Drug: Granulocyte Colony-Stimulating Factor
- Control group
  Interventions: Other: placebo

INTERVENTIONS:
Drug: Granulocyte Colony-Stimulating Factor — Granulocyte-colony stimulating factors (G-CSF) is synthesized in the reproductive tract naturally, it is a hematopoietic lineage-specific cytokine which is known for its specific effects on the activation of intracellular signaling pathways that are associated with the cell proliferation, differentiation, and stimulation of hematopoietic cells of the neutrophilic granulocyte lineage; which act on macrophages of decidual cells and finally affect implantation
  Other Names: filgrastim
  Groups: Intervention group
Other: placebo — mock test without injection of G-CSF
  Groups: Control group

SUMMARY:
Intrauterine infusion of granulocyte colony stimulating factor and reproductive outcomes in infertile women with history of recurrent implantation failure

DETAILED DESCRIPTION:
* Despite the developments in fertility treatment protocols, repeated implantation failure (RIF) still remains a challenging problem for patients and clinicians, it causes deep impact on the quality of life and financial burden, because the majority of failed invitro fertilization- embryo transfer (IVF-ET) cycles exhibit lack of implantation, endometrial receptivity is the limiting factor for implantation and success of IVF programs. Repeated implantation failure (RIF) is defined as pregnancy failure after 2-6 times with at least 10 high quality embryos transferred into the uterus.
* Granulocyte-colony stimulating factors (G-CSF) is synthesized in the reproductive tract naturally, it is a hematopoietic lineage-specific cytokine which is known for its specific effects on the activation of intracellular signaling pathways that are associated with the cell proliferation, differentiation, and stimulation of hematopoietic cells of the neutrophilic granulocyte lineage; which act on macrophages of decidual cells and finally affect implantation.
* During the maturation of the pre-ovulatory follicle, G-CSF receptor expression increases; this also takes place in human endometrium and luteinized granulosa cells. G-CSF receptors also exist on the trophoblast with the highest G-CSF receptor expression occurs in the first trimester. G-CSF effect on recruitment of type 2 T helper cytokine secretion, activation of T regulatory cells, modulation of uterine natural killer and dendritic cells cytotoxicity, as well as endometrium angiogenesis as a result has an essential role on early cross talk between embryo and uterine endometrium. G-CSF stimulates the proliferation and differentiation of endometrial cells by CAMP increase in stromal cell through paracrine and autocrine signaling pathway.
* Studies showed that elevated G-CSF concentrations on follicular fluid increased implantation rate and can improve IVF outcome, it increase the proportion of embryos that develop to the blastocyst stage from 30-76%. Also G-CSF supplemented to the embryo culture medium improves implantation rate. G-CSF can be effective treatment in patient with history of implantation failure and can improve endometrium growth. Also G-CSF may increase pregnancy rate especially in women with thin endometrium.
* In a recent well-designed trial on patients with thin endometrium in which embryo transfer was cancelled with G-CSF treatment in subsequent frozen embryo transfer (FET) cycles, significantly higher implantation rate (31.5% versus 13.9%, P < .01) and clinical pregnancy rate (48.1% vs. 25%, P < .01) was found in those treated with G-CSF in comparison with controls but live birth rate was not statistically significant (33.3% vs. 17.3%).
* In a recent meta-analysis, it was found that the use of G-CSF was associated with significantly higher biochemical (RR 2.385 95% CI:1.414, 4.023) and clinical pregnancy rates (RR 2.312, 95% CI: 1.444, 3.701) among women with thin endometrium or repeated IVF failures in the general population when compared with no treatment or placebos.
* In one of two recent trials with similar patient selection and disease condition, 0.5 ml (300 µg/ml) G-CSF infusion intrauterine at the day of ovum pickup followed by grade A embryo transfer at day 3 was associated with significantly higher pregnancy and implantation rate. 3In the other trial however, the treated group received the same dose of G-CSF subcutaneously 30 min before blastocyst embryo transfer at day 5, there was higher clinical pregnancy, live birth rate and lower abortion rate; but all were not statistically significant.
* This study evaluates the effects of the single dose G-CSF intrauterine infusion in a group of patients with unexplained RIFs 3 days before ET of good quality embryos.

ELIGIBILITY:
Inclusion Criteria:

1. Age group (18-38)
2. History of at least 2 previous IVF or ICSI trial failures with ET of at least 2 good quality embryos in each trial.
3. Endometrial cavity within normal anatomy as assessed with transvaginal ultrasound (TV-US) with or without hysteroscopy and HSG if needed.
4. Availability of good quality embryos (at least 2 grade A embryos) for ET in the investigated trial

Exclusion Criteria:

Any factor which may affect quality of embryos transferred or endometrial receptivity and embryo growth, like:

1. Severe male factor infertility
2. Poor ovarian reserve (according to ESHRE criteria) 1
3. Uterine anatomic factor (eg polyp, intramural fibroid, endometrial septum, intrauterine synechiae .. etc) as well as endometritis
4. Immunological disorder (eg: SLE, APS, … etc)
5. Thyroid or adrenal dysfunction
6. Thrombophilia history or tendency as proven by labs in suspected women
7. Untreated hyperprolactinemia
8. Genetic abnormalities in the infertile couple
9. Chronic hematologic, renal or liver disease

Ages: 18 Years to 38 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Study Population: Infertility patients undergoing ICSI trials at Cairo university school of Medicine IVF unit.
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2024-08-30 (Actual); Study Completion 2024-09-25 (Actual)

PRIMARY OUTCOMES:
Clinical pregnancy rate | 4 weeks after ET
  (GS with viable embryo 4 weeks after ET)

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo university Kasr Alainy OBGYN hospital, Cairo, AlQuahira, Egypt

REFERENCES:
- [Background] Ferraretti AP, La Marca A, Fauser BC, Tarlatzis B, Nargund G, Gianaroli L; ESHRE working group on Poor Ovarian Response Definition. ESHRE consensus on the definition of 'poor response' to ovarian stimulation for in vitro fertilization: the Bologna criteria. Hum Reprod. 2011 Jul;26(7):1616-24. doi: 10.1093/humrep/der092. Epub 2011 Apr 19. PMID 21505041
- [Background] Bashiri A, Halper KI, Orvieto R. Recurrent Implantation Failure-update overview on etiology, diagnosis, treatment and future directions. Reprod Biol Endocrinol. 2018 Dec 5;16(1):121. doi: 10.1186/s12958-018-0414-2. PMID 30518389
- [Background] Eftekhar M, Miraj S, Farid Mojtahedi M, Neghab N. Efficacy of Intrauterine infusion of granulocyte colony stimulating factor on patients with history of implantation failure: A randomized control trial. Int J Reprod Biomed. 2016 Nov;14(11):687-690. PMID 27981253
- [Background] Reda A, Hamid AS, Mostafa R, Refaei E. Comparison between findings of saline infusion sonohysterography and office hysteroscopy in patients with recurrent implantation failure. J Hum Reprod Sci. 2016 Oct-Dec;9(4):236-240. doi: 10.4103/0974-1208.197661. PMID 28216911
- [Background] Arefi S, Fazeli E, Esfahani M, Borhani N, Yamini N, Hosseini A, Farifteh F. Granulocyte-colony stimulating factor may improve pregnancy outcome in patients with history of unexplained recurrent implantation failure: An RCT. Int J Reprod Biomed. 2018 May;16(5):299-304. PMID 30027145
- [Background] Kahyaoglu I, Yilmaz N, Timur H, Inal HA, Erkaya S. Granulocyte colony-stimulating factor: A relation between serum and follicular fluid levels and in-vitro fertilization outcome in patients with polycystic ovary syndrome. Cytokine. 2015 Jul;74(1):113-6. doi: 10.1016/j.cyto.2014.09.002. Epub 2014 Sep 23. PMID 25258001
- [Background] Sugita K, Hayakawa S, Karasaki-Suzuki M, Hagiwara H, Chishima F, Aleemuzaman S, Li JA, Nishinarita S, Yamamoto T. Granulocyte colony stimulation factor (G-CSF) suppresses interleukin (IL)-12 and/or IL-2 induced interferon (IFN)-gamma production and cytotoxicity of decidual mononuclear cells. Am J Reprod Immunol. 2003 Jul;50(1):83-9. doi: 10.1034/j.1600-0897.2003.00024.x. PMID 14506932
- [Background] Rahmati M, Petitbarat M, Dubanchet S, Bensussan A, Chaouat G, Ledee N. Colony Stimulating Factors 1, 2, 3 and early pregnancy steps: from bench to bedside. J Reprod Immunol. 2015 Jun;109:1-6. doi: 10.1016/j.jri.2015.01.005. Epub 2015 Feb 11. PMID 25721620
- [Background] Meier P, Gloekler S, Oezdemir B, Indermuehle A, Traupe T, Vogel R, de Marchi S, Seiler C. G-CSF induced arteriogenesis in humans: molecular insights into a randomized controlled trial. Curr Vasc Pharmacol. 2013 Jan;11(1):38-46. PMID 23391421
- [Background] Gleicher N, Vidali A, Barad DH. Successful treatment of unresponsive thin endometrium. Fertil Steril. 2011 May;95(6):2123.e13-7. doi: 10.1016/j.fertnstert.2011.01.143. Epub 2011 Feb 16. PMID 21324451
- [Background] Gleicher N, Kim A, Michaeli T, Lee HJ, Shohat-Tal A, Lazzaroni E, Barad DH. A pilot cohort study of granulocyte colony-stimulating factor in the treatment of unresponsive thin endometrium resistant to standard therapies. Hum Reprod. 2013 Jan;28(1):172-7. doi: 10.1093/humrep/des370. Epub 2012 Oct 18. PMID 23081869
- [Background] Xu B, Zhang Q, Hao J, Xu D, Li Y. Two protocols to treat thin endometrium with granulocyte colony-stimulating factor during frozen embryo transfer cycles. Reprod Biomed Online. 2015 Apr;30(4):349-58. doi: 10.1016/j.rbmo.2014.12.006. Epub 2014 Dec 30. PMID 25682303
- [Background] Li J, Mo S, Chen Y. The effect of G-CSF on infertile women undergoing IVF treatment: A meta-analysis. Syst Biol Reprod Med. 2017 Aug;63(4):239-247. doi: 10.1080/19396368.2017.1287225. Epub 2017 Feb 28. PMID 28632452
- [Derived] Elkhateb I, Fahmy R, Ramadan W, Mourad A, El-Demiry NM, Shohayeb A. Granulocyte colony-stimulating factor for recurrent implantation failure: the results of a 5-years cohort study. Sci Rep. 2025 Nov 18;15(1):40390. doi: 10.1038/s41598-025-24587-3. PMID 41254175